CLINICAL TRIAL: NCT01118741
Title: A Multi-institutional Translational Clinical Trial of Disulfiram in Men With Recurrent Prostate Cancer as Evident by a Rising PSA
Brief Title: Study of Recurrent Prostate Cancer With Rising Prostate Specific Antigen (PSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0972
Record Dates: First submitted 2010-04-29; First posted 2010-05-07 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Rising PSA; Recurrent Non Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Disulfiram — Cohort 1: 250mg PO daily for 28 days Cohort 2: 500mg PO daily for 28 days
  Other Names: Antabuse

SUMMARY:
disulfiram is a DNA methyltransferase inhibitor that may provide benefit for patients with prostate cancer by restoring tumor suppressor genes.

DETAILED DESCRIPTION:
The primary hypothesis of this study is that disulfiram is a DNA methyltransferase inhibitor and may provide benefit for patients with prostate cancer by restoration of tumor suppressor genes. Disulfiram is a potent DNA methyltransferase 1 (DNMT1) inhibitor in vitro in our laboratory and it was recently found as one of the most potent inhibitors for PCa growth in vitro by screening the Johns Hopkins Drug Library. Based on this data, extensive in vitro and in vivo studies have been performed to explore its potential antitumor activities in prostate PCa. Using both androgen sensitive and insensitive PCa cell lines, we have confirmed that disulfiram can demethylate known highly methylated tumor suppressor genes such as APC and RARß in PCa cell lines. Disulfiram inhibited PCa cell growth in vitro and in vivo. In addition to these new findings, the antitumor activity of disulfiram and its other possible mechanisms of action are well documented in literature. Disulfiram has been shown to induce apoptosis in a number of cell lines including PCa. A variety of underlying mechanisms of anticancer activity have been reported. Disulfiram has been shown to reduce angiogenesis, inhibit DNA topoisomerases, inhibit nuclear factor κB, induce p21 and p53 with G1/S cell cycle arrest, induce pro-apoptotic redox-related mitochondrial membrane permeabilization, inactivate Cu/Zn superoxide dismutase by Cu2+ complexation, inhibit Zn2+-dependent matrix metalloproteinases, and prevent tumor invasion or metastasis. The disulfiram analogue pyrrolidine dithiocarbamate (PDTC) has been shown to inhibit proteasomal activity in combination with copper in human breast and PCa cell lines. Also, disulfiram or its metabolites permanently inactivate the human multidrug resistance P-glycoprotein or reverses either MDR1- or MRP1-mediated drug efflux.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and HIPAA authorization for the release of personal health information.
* Adult male ≥18 years of age
* No desire to drink any alcohol during the study period. (The potential for ethanol interactions may last 7 to 14 days. Patient is allowed to drink alcohol 2 weeks after the study is finished)
* Histological confirmed diagnosis of adenocarcinoma of the prostate (M0) with evidence of biochemical relapse after local therapy (i.e., surgery, radiation therapy, or both). Baseline PSA must be ≥ 1 ng/ml.
* There must be a confirmed rise in PSA shown by 2 PSA values at least 1 week apart, higher than a reference value noted within 12 months of study entry. Interim PSA values during the immediate pre-study 12-month interval may demonstrate a "fluctuation" including a decline; however the study baseline PSA must have show a rise within the pre-study 12-months period. Baseline PSA must be determined within 4 weeks of study entry. At least 3 PSA values are necessary to calculate PSA doubling time via PSADT calculator.
* All previous local modalities of treatment, including radiation and surgery, must have been discontinued at least 4 weeks prior to treatment in this study. Patients may have received prior systemic chemotherapy, hormonal therapy, biologic or vaccine therapy
* Patients receiving intermittent hormonal therapy for their rising PSA state are considered eligible if testosterone level is above 150ng/dl and treatment was discontinued > 6 months and agree not to have additional injections while on study drug.
* No history of or current clinical or radiological evidence of distant metastases (excluding prostascint scan/PET in absence of radiographic disease in Bone scan, CT scan or MRI if used). Retroperitoneal/pelvic lymph node up to 2 cm size is allowed for the study.
* ECOG performance score < 2 within 14 days before being registered for protocol therapy
* Normal organ function with acceptable initial laboratory values:

  * Absolute neutrophil count ≥ 1 x 109/L
  * Platelets > 50 x 109/L
  * Creatinine <2 mg/dL
  * Bilirubin <1.5 X ULN (institutional upper limits of normal)
  * AST (SGOT) and ALT (SGPT) ≤ 1.5 x ULN
  * Willingness to use adequate methods of contraception throughout study participation and for at least 3 months after completing therapy

Exclusion Criteria:

* Metastatic disease or currently active second malignancy
* History of alcohol dependence, seizures or psychoses.
* Medical conditions such as uncontrolled hypertension, uncontrolled diabetes mellitus, cardiac disease, active infectious hepatitis, type A, B or C, hypothyroidism, which would, in the opinion of the investigator, make this protocol unreasonably hazardous
* Major thoracic or abdominal surgery within the prior 3 weeks. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* Use of any prohibited concomitant medications: Metronidazole, Amprenavir, Paraldehyde, Phenytoin, Coumadin, alcohol or alcohol-containing preparations, Isoniazid, Amitriptyline (please see Appendix B for other potential drug-drug interactions). The washout period is at least 2 weeks before starting the study
* Insufficient time from last prior regimen or radiation exposure: Systemic therapies for prostate cancer within 28 days prior to disulfiram; strontium-89 within 12 weeks; bicalutamide within 6 weeks.
* Persistent Grade >2 treatment-related toxicity from prior therapy
* History of any disulfiram-related or drug induced anaphylactic reaction
* Receipt of another investigational agent within 28 days of study entry. Patient must have recovered from all side effects of prior investigational therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Carducci, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - Thomas Jefferson Universith, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: 06/04/2010 through 08/01/2011 in medical clinics
Pre-assignment Details: Given the toxic effects of disulfiram when administered within 14 days of ingesting ethanol, participants were required to agree not to drink alcohol during the study and for 14 days after its completion.
Groups:
- Disulfiram Low Dose 250mg Dose: First 9 subjects were assigned to the low dose (250mg) arm. These subjects took 250mg daily for 28 days per cycle.
- Disulfiram High Dose 500mg Dose: After accrual to the low dose was complete,ten subjects were assigned to the high dose (500mg) arm. These subjects took 500mg daily for 28 days per cycle.
Period: Overall Study
Arm/Group | Disulfiram Low Dose 250mg Dose | Disulfiram High Dose 500mg Dose
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Disulfiram Low Dose 250mg Dose: First 9 subjects were assigned to the low dose arm
- Disulfiram High Dose 500mg Dose: After 9 subjects were enrolled in the low dose arm, the high dose was opened.
- Total: Total of all reporting groups
Arm/Group | Disulfiram Low Dose 250mg Dose | Disulfiram High Dose 500mg Dose | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 11
  >=65 years | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (7.0) | 62.6 (3.4) | 64.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a Demethylation Response at Each Dose Level
Description: For both of the doses explored (i.e. disulfiram 250 mg PO daily and 500 mg PO daily) the proportion of subjects with a demethylation response was computed. A demethylation response was defined as a >=10% decrease from baseline in global 5-methyl cytosine content as assessed from peripheral blood mononuclear cells.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Disulfiram Low Dose 250mg Dose | Disulfiram High Dose 500mg Dose
Number analyzed (Participants) | 9 | 10
proportion of participants | .22 [0.03 to 0.60] | .30 [0.07 to 0.65]

2. Secondary Outcome: Clinical Response
Description: To assess the clinical response measured by prostate specific antigen (PSA) progression at 6 months after treatment with the defined dose of disulfiram in prostate cancer (PCa) patients with evidence of biochemical relapse after local therapy. Reported as number of participants with PSA progression by 6 months.
  Criteria used to assess: A rise in PSA noted at 6 months, greater than 50% over PSA value at baseline and > 2 ng/ml, above the nadir. The rise was confirmed by a second PSA value obtained at least 1 week from that reference value.
Time Frame: Up to 6 months
Measure: Number; unit: participants
Arm/Group | Disulfiram Low Dose 250mg Dose | Disulfiram High Dose 500mg Dose
Number analyzed (Participants) | 9 | 10
participants | 5 | 0

ADVERSE EVENTS:
Time Frame: 7/16/10-9/27/11 (14 months)
Arm/Group | Disulfiram Low Dose 250mg Dose | Disulfiram High Dose 500mg Dose
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 6/9 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disulfiram Low Dose 250mg Dose (N=9) | Disulfiram High Dose 500mg Dose (N=10)
FATIGUE (General disorders) | 6 (6) | 8 (8)
HEARING LOSS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TASTE ALTERATION (Gastrointestinal disorders) | 2 (2) | 4 (4)
DIPLOPIA (Eye disorders) | 1 (1) | 0 (0)
ALT (Investigations) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No